CLINICAL TRIAL: NCT04061161
Title: Anti-inflammatory Effects of Tiotropium in Patients with Stable COPD- a Multicenter Randomized Controlled Double-blind Study
Brief Title: Anti-inflammatory Effects of Tiotropium in Patients with Stable COPD
Acronym: ANTIOFLAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Huib A.M. Kerstjens, Full professor pulmonology; Head of department of Pulmonology and Tuberculosis; Principal Investigator, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-002173-22
Record Dates: First submitted 2019-08-14; First posted 2019-08-19 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2023-08

CONDITIONS: COPD
Keywords: Tiotropium; Anti-inflammatory effects; TNF-alpha mRNA in induced sputum
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Intervention Model Description: This will be a multicenter parallel design randomized placebo controlled double-blinded study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tiotropium respimat (Active Comparator): Tiotropium respimat 2.5mcg two actuations once daily
  Interventions: Drug: Tiotropium Bromide
- Placebo respimat (Placebo Comparator): Placebo respimat two actuations once daily
  Interventions: Drug: Tiotropium Bromide

INTERVENTIONS:
Drug: Tiotropium Bromide — Participants will be double-blind randomized for Tiotropium or Placebo treatment for 6 weeks

SUMMARY:
This study aims to assess the anti-inflammatory effects after 6 weeks treatment with tiotropium compared to placebo in patients with stable COPD

DETAILED DESCRIPTION:
Rationale: Acetylcholine is the primary parasympathetic neurotransmitter in the airways, and induces bronchoconstriction. Since the cholinergic tone appears to be the major reversible component of obstruction, muscarinic receptor antagonism and bronchodilation represent the primary goal of anticholinergic therapy in patients with chronic obstructive pulmonary disease (COPD). Long-acting anticholinergic therapy is central in GOLD stage B-D, because of improvements in lung function, quality of life, and especially reduction of exacerbations. The elicited reduction in exacerbations with the long-acting muscarinic antagonist (LAMA) tiotropium appears larger than that of the long-acting beta agonist (LABA) salmeterol even when the bronchodilation is similar. In asthma too, it has been shown that the addition of the tiotropium to inhaled corticosteroids (ICS)+LABA combination therapy reduces the number of severe exacerbations. These effects on exacerbation frequency suggest that tiotropium might exert anti-inflammatory effects in the airways next to bronchodilatory effects. There are multiple animal and in vivo studies to indeed suggest an anti-inflammatory effect of anticholinergics.

Such an anti-inflammatory effect of anticholinergic intervention could be clinically relevant; however it has not been previously demonstrated in patients with COPD.

The investigators hypothesize that tiotropium bromide reduces the ongoing inflammation in patients with COPD compared to placebo. The investigators expect a decrease of TNF-alpha mRNA in sputum after treatment with tiotropium bromide.

Objective: This research proposal aims to assess the anti-inflammatory effects after 6 weeks treatment with tiotropium compared to placebo in patients with stable COPD.

Study design: This will be a multicenter parallel design randomized controlled double-blinded study.

Study population: A total of 50 COPD patients with stable disease status will be included and followed for two consecutive visits.

Intervention: COPD patients will be randomized to the treatment group (tiotropium respimat 5 ug) or to the placebo group.

Main study parameters/endpoints: A decrease of TNF-alpha mRNA in induced sputum will be the main parameter for assessing the anti-inflammatory effects of 6 week treatment with tiotropium in patients with stable COPD. Additionally, changes in sputum cell differentials and other cytokine parameters (protein, mRNA,LTB4), blood cell differentials, CRP, and cytokine parameters, health related quality of life (CCQ, CAT) will be assessed as well as changes in post-bronchdilator FEV1.

ELIGIBILITY:
Inclusion Criteria:

* • Men or women, age >= 40 years.

  * A diagnosis of COPD according to the criteria of the GOLD organization
  * Post-bronchodilator FEV1 / FVC ratio < 70% (ERS equations) and post-bronchodilator FEV1 < 80%pred.
  * A smoking history of > 10 pack years.
  * post-bronchodilator FEV1 > 1.5 Litres and ability to produce sputum after hypertonic saline induction.
  * No upper or lower respiratory tract infection in the last 4 weeks necessitating antibiotic treatment or consisting of quite probable viral etiology.
  * Being in a stable phase of COPD, as judged by the investigator. No courses of systemic steroids or antibiotics for respiratory problems last 4 weeks
  * The participant needs to be able to understand the Dutch language
  * Signed and dated informed consent obtained before any study related procedures (including withdrawal of concomitant medication) are conducted.

Exclusion Criteria:

* • Treatment with immune-modulating agents for any disease, including leuktriene receptor antagonists,

  * Treatment with long-acting anticholinergics <4 weeks before the start of the study.
  * Treatment with corticosteroids <4 weeks before the start of the study.
  * Targeted lung denervation therapy in the past.
  * Concomitant diagnosis of asthma.
  * Any significant other pulmonary disease or disorder (e.g. known alpha1-antitrypsine deficiency, significant bronchiectasis), as judged by the investigator.
  * Narrow angle glaucoma.
  * Azithromycine maintenance treatment.
  * Active malignant disease (at least 5 years malignant disease-free)
  * Other significant disease or disorder (like cardiovascular, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic (including diagnosed diabetes), malignant, psychiatric, major physical impairment), which, in the opinion of the investigators may either put the patient at risk because of participation in the study, or may influence the results of the study, or the patient's ability to participate in the study.
  * Females of childbearing potential without an efficient contraception unless they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH >40 mIU/mL or the use of one or more of the following acceptable methods of contraception:

    1. Surgical sterilization (e.g. bilateral tubal ligation, hysterectomy).
    2. Hormonal contraception (implantable, patch, oral, injectable).
    3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/cream/suppository.
    4. Continuous abstinence.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in concentration of TNF-alpha (mRNA level) in induced sputum | 6 week treatment duration
  To assess whether 6 weeks treatment with tiotropium elicts anti-inflammatory effects compared to placebo in patients with stable COPD, as measured by a change in TNF-alpha mRNA level in induced sputum

SECONDARY OUTCOMES:
Change in concentration of sputum cell differentials in induced sputum | 6 week treatment duration
  To assess whether 6 weeks treatment with tiotropium elicts anti-inflammatory effects compared to placebo in patients with stable COPD, as measured by a change in sputum cell differentials (% of total cells) in induced sputum
Change in concentration of LTB4 level in induced sputum | 6 week treatment duration
  To assess whether 6 weeks treatment with tiotropium elicts anti-inflammatory effects compared to placebo in patients with stable COPD, as measured by a change in LTB4 level (pg/ml) in induced sputum
Change in concentration of cytokine protein level in induced sputum | 6 week treatment duration
  To assess whether 6 weeks treatment with tiotropium elicts anti-inflammatory effects compared to placebo in patients with stable COPD, as measured by a change in cytokine protein levels (IL-8,IL-6,MCP-1, TNF-a, MIP-1beta,TGF-beta,MPO, ECP; pg/ml) in induced sputum
Change in concentration of cytokine mRNA level in induced sputum | 6 week treatment duration
  To assess whether 6 weeks treatment with tiotropium elicts anti-inflammatory effects compared to placebo in patients with stable COPD, as measured by a change in cytokine mRNA levels of IL-8,IL-6,MCP-1, TNF-a, MIP-1beta,TGF-beta,MPO, ECP in induced sputum
Change in concentration of cell differentials + CRP in blood serum | 6 week treatment duration
  To assess whether 6 weeks treatment with tiotropium elicts anti-inflammatory effects compared to placebo in patients with stable COPD, as measured by a change in cell differentials (10^9/L) +CRP (mg/L) in blood serum
Change in concentration cytokine protein level in blood serum | 6 week treatment duration
  To assess whether 6 weeks treatment with tiotropium elicts anti-inflammatory effects compared to placebo in patients with stable COPD, as measured by a change in cytokine protein levels (IL-6,TNF-a,siCAM; pg/ml) in blood serum
Change in health related quality of life (CCQ, CAT questionnaires) | 6 week treatment duration
  To assess whether 6 weeks treatment with tiotropium elicts anti-inflammatory effects compared to placebo in patients with stable COPD, as measured by a changein health related quality of life (CCQ and CAT questionnaires)

OTHER OUTCOMES:
Differences in gene expression measured in sputum samples | 6 week treatment duration
  RNA-sequencing of sputum samples

CONTACTS AND LOCATIONS:
Overall Officials: Wouter van Geffen, MD PhD, Principal Investigator — Medical centrum Leeuwarden, Department of pulmonology
Locations (2):
- Netherlands (2):
  - University Medical Center, Groningen
  - Medical centrum Leeuwarden, Leeuwarden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bathoorn E, Liesker J, Postma D, Koeter G, van Oosterhout AJ, Kerstjens HA. Safety of sputum induction during exacerbations of COPD. Chest. 2007 Feb;131(2):432-8. doi: 10.1378/chest.06-2216. PMID 17296644
- [Background] Brightling CE, Monterio W, Green RH, Parker D, Morgan MD, Wardlaw AJ, Pavord D. Induced sputum and other outcome measures in chronic obstructive pulmonary disease: safety and repeatability. Respir Med. 2001 Dec;95(12):999-1002. doi: 10.1053/rmed.2001.1195. PMID 11778799
- [Background] Gosens R, Zaagsma J, Meurs H, Halayko AJ. Muscarinic receptor signaling in the pathophysiology of asthma and COPD. Respir Res. 2006 May 9;7(1):73. doi: 10.1186/1465-9921-7-73. PMID 16684353
- [Background] Kerstjens HA, Engel M, Dahl R, Paggiaro P, Beck E, Vandewalker M, Sigmund R, Seibold W, Moroni-Zentgraf P, Bateman ED. Tiotropium in asthma poorly controlled with standard combination therapy. N Engl J Med. 2012 Sep 27;367(13):1198-207. doi: 10.1056/NEJMoa1208606. Epub 2012 Sep 2. PMID 22938706
- [Background] Kistemaker LE, Bos IS, Menzen MH, Maarsingh H, Meurs H, Gosens R. Combination therapy of tiotropium and ciclesonide attenuates airway inflammation and remodeling in a guinea pig model of chronic asthma. Respir Res. 2016 Feb 4;17:13. doi: 10.1186/s12931-016-0327-6. PMID 26846267
- [Background] Kistemaker LE, Gosens R. Acetylcholine beyond bronchoconstriction: roles in inflammation and remodeling. Trends Pharmacol Sci. 2015 Mar;36(3):164-71. doi: 10.1016/j.tips.2014.11.005. Epub 2014 Dec 13. PMID 25511176
- [Background] Kistemaker LE, Oenema TA, Meurs H, Gosens R. Regulation of airway inflammation and remodeling by muscarinic receptors: perspectives on anticholinergic therapy in asthma and COPD. Life Sci. 2012 Nov 27;91(21-22):1126-33. doi: 10.1016/j.lfs.2012.02.021. Epub 2012 Mar 3. PMID 22406302
- [Background] Perng DW, Tao CW, Su KC, Tsai CC, Liu LY, Lee YC. Anti-inflammatory effects of salmeterol/fluticasone, tiotropium/fluticasone or tiotropium in COPD. Eur Respir J. 2009 Apr;33(4):778-84. doi: 10.1183/09031936.00115308. Epub 2009 Jan 7. PMID 19129278
- [Background] Powrie DJ, Wilkinson TM, Donaldson GC, Jones P, Scrine K, Viel K, Kesten S, Wedzicha JA. Effect of tiotropium on sputum and serum inflammatory markers and exacerbations in COPD. Eur Respir J. 2007 Sep;30(3):472-8. doi: 10.1183/09031936.00023907. Epub 2007 May 15. PMID 17504798
- [Background] Tashkin DP, Celli B, Senn S, Burkhart D, Kesten S, Menjoge S, Decramer M; UPLIFT Study Investigators. A 4-year trial of tiotropium in chronic obstructive pulmonary disease. N Engl J Med. 2008 Oct 9;359(15):1543-54. doi: 10.1056/NEJMoa0805800. Epub 2008 Oct 5. PMID 18836213
- [Background] "Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report: GOLD Executive Summary." Claus F. Vogelmeier, Gerard J. Criner, Fernando J. Martinez, Antonio Anzueto, Peter J. Barnes, Jean Bourbeau, Bartolome R. Celli, Rongchang Chen, Marc Decramer, Leonardo M. Fabbri, Peter Frith, David M.G. Halpin, M. Victorina Lopez Varela, Masaharu Nishimura, Nicolas Roche, Roberto Rodriguez-Roisin, Don D. Sin, Dave Singh, Robert Stockley, Jorgen Vestbo, Jadwiga A. Wedzicha and Alvar Agusti. Eur Respir J 2017; 49: 1700214. Eur Respir J. 2017 Jun 22;49(6):1750214. doi: 10.1183/13993003.50214-2017. Print 2017 Jun. No abstract available. PMID 28642306
- [Background] Vogelmeier C, Hederer B, Glaab T, Schmidt H, Rutten-van Molken MP, Beeh KM, Rabe KF, Fabbri LM; POET-COPD Investigators. Tiotropium versus salmeterol for the prevention of exacerbations of COPD. N Engl J Med. 2011 Mar 24;364(12):1093-1103. doi: 10.1056/NEJMoa1008378. PMID 21428765